CLINICAL TRIAL: NCT06509646
Title: Comparison of Tai Chi and Frenkel's Exercises to Improve Balance, Fall Risk and Activities of Daily Living in Patients With Stroke
Brief Title: Comparison of Tai Chi and Frenkel's Exercises in Patients With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0285 Faraha
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: Tai Chi Exercise; Frenkel's Exercise; Stroke; ADL; Fall Risk; Balance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single blinded as assessor of the study would be kept blind of the treatment groups to which patient will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goup A (Tia Chi Exercise) (Experimental): * Warm up 5 minutes
  * Routine Physical Therapy 20 minutes (which may include exercises such as stretching, strengthening, and range-of- motion exercises)
  * Rest Interval 5 minute
  * Yang style 24-posture short-form (16) for 30 minute Intensity: low Frequency: 1-2 times/week. Duration: ≤30 min (minutes)(18)
  * Cool down 5 mins.
  Interventions: Other: Tia Chi Exercise
- Group B (Frenkel's Exercise ) (Active Comparator): * Warm up 5 minutes
  * Routine Physical Therapy 20 minutes (which may include exercises such as stretching, strengthening, and range-of- motion exercises)
  * Rest Interval 5 minute
  * Frenkel's exercises 30 minutes (Through these exercises, the patients would learn how to stay balanced and prevent falls by using their visual, somatosensory, and vestibular systems) 4. Rest interval 5 minutes 5. Intensity: low 6. Frequency: 1-2 times/week. 7. Duration: ≤30 min (minutes) 8. Cool down 5 mins
  Interventions: Other: Frenkel's Exercise

INTERVENTIONS:
Other: Tia Chi Exercise — • Yang style 24-posture short-form (16) for 30 minute It consists of 24 unique movements that are performed in a sequence. The form is designed to be easy to learn and can be completed in about six minutes.
  Treatment dosage will be 1 session per day of 1 hour class, 2 sets per session, and 5 repetitions per set, 3 times per week and for 12 weeks
  Arms: Goup A (Tia Chi Exercise)
Other: Frenkel's Exercise — Frenkel's exercises 30 minutes (Through these exercises, the patients would learn how to stay balanced and prevent falls by using their visual, somatosensory, and vestibular systems).
  Treatment dosage will be 1 session per day of 1 hour class, 2 sets per session, and 5 repetitions per set, 3 times per week and for 12 weeks
  Arms: Group B (Frenkel's Exercise )

SUMMARY:
The main objective of this study is to compare the effectiveness of Tai Chi and Frenkel's exercises to improve balance, fall risk and activities of daily living in patients with stroke.

DETAILED DESCRIPTION:
A total of 44 patients will be recruited after inclusion and exclusion criteria. Patients will be recruited through nonprobability convenience sampling technique and will be randomized through Lottery method into either a Group A or a Group B, and for each group, the number of patients will be identical. Group A will receive Tai Chi exercises for 1-hour class, 3 times per week for 12 weeks along with routine physical therapy. Routine treatment includes range of motion (ROM) exercise, stretching & strengthening exercises, passive movements & gait training. Group A will receive the Tai Chi exercise with conventional treatment and Group B will receive Frenkel's exercise with conventional treatment. Treatment dosage will be 1 session per day of 1 hour class, 2 sets per session, and 5 repetitions per set, 3 times per week and for 12 weeks. Patients will be assessed at baseline and after the treatment using a variety of measurement scales. After the completion of this time period, the assessment of balance, activities of daily living and fall risk will be performed again and will be compared to baseline assessment to check the comparison between 2 interventions. The risk fall will be measured by Stratify Risk Assessment Tool, Activities of daily will be measured by The Barthel Index (BI) , while balance will be assessed by using berg balance scale (BBC). Data will be analyzed by using SPSS (Statistical Package for Social Sciences) 23 version.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling survivors of stroke who were aged ≥50 years
* Both genders can participate in the study
* ≥3 months poststroke
* The vital signs were stable
* Survivors of both hemorrhagic and ischemic stroke
* Modified Rankin Scale 14 score of three or less
* Short Physical Performance Battery 15 score of 3 to 9
* Mini-Mental State Exam 16,17 score of 18 or greater.

Exclusion Criteria:

* The subject is unable to perform exercises.
* Subjects with diagnosed vestibular disease.
* The subjects included in the experiment were normal elderly without stroke diseases.
* The subjects had dyskinesias and could not complete Tai Chi exercises.
* Serious medical condition (e.g. active cancer treatment.
* Stroke survivors whom had no disability that would interfere with study participation.
* Subject taking medications that increases the incidence of fall.
* Subjects who undergoes strength and balance training in the past 3 months.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-12 (Estimated); Study Completion 2024-07-20 (Estimated)

PRIMARY OUTCOMES:
The Barthel Index | 12th week
  The scoring is as follows: 0 = unable, 1 = needs assistance/help, 2 = independent. The for the ten items are summed and x 5 to get a total score out of 100. Proposed guidelines for interpreting Barthel scores are as follows: scores of 0-20 indicate "total" dependency.
The Berg Balance Scale (BBS) | 12th week
  The Berg Balance Score (BBS) is the best-known balance measurement tool, originally designed to measure balance in older individuals. It consists of 14 items scored on an ordinal scale of 0 to 4 for a total of 56 points (a higher score indicates lower fall risk)
Fall Risk Assessment Tool (SRATIFY) | 12th week
  The STRATIFY Scale is a tool used to identify risk factors for falls in hospitalized patients, using a 0-5 score to predict patients who will fall. It consists of five questions that assess the patient's history of falls, agitation, visual impairment, toileting needs, and mobility. The total score may be used to predict future falls, but it is more important to identify risk factors using the scale and then plan care to address those risk factors. The tool has good test-retest reliability and moderate inter-rater reliability

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, phd, Principal Investigator — Riphah International University
Locations (1):
- Alveena fatima, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No